CLINICAL TRIAL: NCT07019753
Title: Experience With the Use of Continuous Glucose Monitoring (CGM) Devices in People With Type 2 Diabetes Mellitus
Acronym: Glucocavi
Status: Not yet recruiting | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Sergi Rodríguez Soler, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: 25/003-P
Record Dates: First submitted 2025-04-26; First posted 2025-06-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Patient Satisfaction; Continuous Glucose Monitoring; Type 2 Diabetes Mellitus (T2DM)
Keywords: Continuous Glucose Monitoring; Patient Satisfaction; Type 2 Diabetes Mellitus (T2DM); Quality of Life; Primary Care
MeSH Terms: conditions — Patient Satisfaction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 2 diabetes and continuous glucose monitoring Tarragona: People with T2DM and intensive insulin therapy who have used a CGM device for at least the last 12 months in the Camp de Tarragona health region.

SUMMARY:
Background: In recent years, diabetes management has evolved with the introduction of continuous glucose monitoring (CGM) devices. Some qualitative studies have been conducted to assess the experiences of patients with type 2 diabetes mellitus (T2DM) using CGM devices, but none have been conducted in a Mediterranean country. Furthermore, there are differences in the amount of time study participants used the CGM device, ranging from 14 days to 6 months, and in some studies, participants did not receive insulin treatment.

Objectives: To understand the benefits and barriers described by people with type 2 diabetes mellitus who use CGM devices through inductive thematic analysis of interviews conducted with them.

Methodology: Qualitative study with a phenomenological approach and conversational technique. Adults with T2DM who have used a CGM device continuously for the past 12 months will be interviewed individually.

Data analysis: They will be analyzed using inductive thematic analysis. The interviews will be transcribed verbatim, along with any relevant data collected by the other researcher present at the interview. Three researchers will then conduct a preliminary analysis, from which codes will be agreed upon and themes, categories, and subcategories will be proposed through triangulation among the researchers. This will be done inductively, through analysis, in-depth reflection, and debate among the three researchers.

Applicability and relevance: Knowing the opinion of people with T2DM who use CGM devices, as well as the barriers and facilitators they find to its use will help healthcare professionals to better understand their patients and thus provide more personalised and closer healthcare. In addition, healthcare managers and administrators will be able to find out whether patients find it useful to use a CGM device, whether they reduce the use of capillary glycaemia strips, whether they become more aware of their disease and increase their self-monitoring, etc. All this will help to decide whether it is beneficial to extend the indication of these devices to more people with type 2 diabetes.

DETAILED DESCRIPTION:
Background: Diabetes mellitus is a chronic disease that affects millions of people worldwide. More than 95% of cases are T2DM. The CGM devices are attached to the skin and allow continuous measurement of glucose levels, monitoring glucose trends, and the rate at which glucose level rise and fall without the need for capillary glycaemias test, making glycemic control easier for people with diabetes.

Study development: The recruitment period runs from January 2026 to April 2026. Opinion sampling will be conducted. Participants will be recruited by health professionals (nurse or doctor) CGM referents from each of the 20 primary care centres in the Camp de Tarragona health region. They will explain the study and will invite all people who meet all the inclusion criteria and none of the exclusion criteria to participate in the study.

The principal investigator will select between 5 and 10 participants from those preselected by the CGM referents, taking into account the sample's diverse profiles: age, gender, years of diabetes evolution, metabolic control, etc.

Interviews will last between 30 and 60 minutes, and interviews will continue until data saturation is reached (anticipated between 5 and 10).

Participants must sign an informed consent and their data will be coded.

Data analysis: In order to facilitate the inductive analysis of the interview data, the ATLAS-TI software (version 8 or later) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Have been using a CGM sensor daily for diabetes management for the past 12 months or more.
* Treatment with intensive insulin therapy (basal bolus regimen with 3 or more daily doses of insulin).
* Agree to participate in the study.

Exclusion Criteria:

* Cognitive impairment measured by the SPMSQ test with a score of 3 or more errors.
* Being institutionalised.
* Have another person responsible for monitoring the device and making decisions related to diabetes (insulin adjustment, carbohydrate rations, etc.).
* Language difficulty: not being able to hold a fluent conversation in Catalan or Spanish for 30-60 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in an industrialised country with a diagnosis of type 2 diabetes with intensive insulin regimen who have used a CGM device for at least the last 12 months. Participants will be recruited from primary care centres in the Camp de Tarragona health region following inclusion and exclusion criteria. Depending on the location of the primary care centre, the population may be from an urban, semi-urban, or rural setting.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Participants' experience | Last 12 months using the CGM device.
  The themes, categories, and subcategories that emerge from the analysis of each interview will be compared with those of the other participants to determine what similarities and contrasts exist.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Rodríguez-Soler, Nurse, Principal Investigator — Institut Català de la Salut
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] Chiu CJ, Chou YH, Chen YJ, Du YF. Impact of New Technologies for Middle-Aged and Older Patients: In-Depth Interviews With Type 2 Diabetes Patients Using Continuous Glucose Monitoring. JMIR Diabetes. 2019 Feb 21;4(1):e10992. doi: 10.2196/10992. PMID 30789351
- [Background] Shin M, Yang Y, Kang JH, Jin HY. Exploring the Initial Encounter with Continuous Glucose Monitoring among Individuals with Type 2 Diabetes: A Two-Week Trip. Diabetes Metab Syndr Obes. 2024 Sep 20;17:3521-3534. doi: 10.2147/DMSO.S466734. eCollection 2024. PMID 39319303
- [Background] Johansson UB, Andreassen Gleissman S, Korkeila Liden M, Wickman M, Gustafsson B, Sjoberg S. Mixed methods study on the feasibility of implementing periodic continuous glucose monitoring among individuals with type 2 diabetes mellitus in a primary care setting. Heliyon. 2024 Apr 16;10(8):e29498. doi: 10.1016/j.heliyon.2024.e29498. eCollection 2024 Apr 30. PMID 38660249
- [Background] Allen NA, Jacelon CS, Chipkin SR. Feasibility and acceptability of continuous glucose monitoring and accelerometer technology in exercising individuals with type 2 diabetes. J Clin Nurs. 2009 Feb;18(3):373-83. doi: 10.1111/j.1365-2702.2008.02533.x. PMID 19191984
- [Background] Sergel-Stringer OT, Wheeler BJ, Styles SE, Boucsein A, Lever CS, Paul RG, Sampson R, Watson A, de Bock MI. Acceptability and experiences of real-time continuous glucose monitoring in adults with type 2 diabetes using insulin: a qualitative study. J Diabetes Metab Disord. 2024 Mar 5;23(1):1163-1171. doi: 10.1007/s40200-024-01403-9. eCollection 2024 Jun. PMID 38932793
- [Background] Hirsch IB. Introduction: History of Glucose Monitoring. In: Role of Continuous Glucose Monitoring in Diabetes Treatment. Arlington (VA): American Diabetes Association; 2018 Aug. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK538968/ PMID 34251770
- [Background] Litchman ML, Allen NA, Sanchez-Birkhead A, Ng A, Rodriguez-Gonzales B, Iacob E, Greenwood DA. Continuous Glucose Monitoring Plus an Online Peer Support Community Reinforces Healthy Behaviors in Hispanic Adults With Type 2 Diabetes. Diabetes Spectr. 2022 Fall;35(4):452-460. doi: 10.2337/ds21-0067. Epub 2022 Mar 28. PMID 36561654